CLINICAL TRIAL: NCT06232629
Title: Towards Noninvasive Deep Brain Stimulation of the Basal Ganglia in Parkinson's Disease Using Low-intensity Transcranial Ultrasound Stimulation
Brief Title: Towards Noninvasive DBS of the Basal Ganglia in Parkinson's Disease Using TUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Robert Chen, Senior Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-5740#4
Record Dates: First submitted 2023-12-26; First posted 2024-01-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Dystonia
Keywords: Transcranial Ultrasound Stimulation; Local Field Potential; Globus Pallidus
MeSH Terms: conditions — Parkinson Disease; Dystonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will be blind to stimulation conditions (sham/active TUS). The assessor will be blind to the stimulation condition (sham/active TUS) while analyzing LFPs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Low-Intensity Transcranial Focused Ultrasound (Active Comparator): NeuroFUS device stimulation with 4-channel transducer Stimulation target = GPi Stimulation parameters = 5Hz and 10 Hz protocols at ISPPA=30 W/cm2
  Interventions: Device: TUS Active
- Sham Low-Intensity Transcranial Focused Ultrasound (Sham Comparator): NeuroFUS device stimulation with 4-channel transducer Stimulation target = GPi and occipital cortex Stimulation parameters = for the passive sham protocol: GPi target (5Hz and 10 Hz protocols at 0 ISPPA) and for the active sham protocol: occipital target (5Hz and 10 Hz protocol at 30 ISPPA)
  Interventions: Device: TUS Sham

INTERVENTIONS:
Device: TUS Active — Bilateral GPis will be sonicated using NeuroFUS device for either two minutes (5Hz protocol) or 40 seconds (10 Hz protocol) per hemisphere and with 30 W/cm2 Isppa
  Arms: Active Low-Intensity Transcranial Focused Ultrasound
Device: TUS Sham — Passive sham: Bilateral GPis will be sonicated using NeuroFUS device for two minutes (5Hz protocol) or 40 seconds (10 Hz protocol) per hemisphere and 0 W/cm2 Isppa
  Active sham: Bilateral occipital cortices will be sonicated using NeuroFUS device for two minutes (5Hz protocol) or 40 seconds (10 Hz protocol) per hemisphere and 30 W/cm2 Isppa
  Arms: Sham Low-Intensity Transcranial Focused Ultrasound

SUMMARY:
Transcranial Ultrasound Stimulation (TUS) is an emerging non-invasive brain stimulation technique capable of targeting both superficial and deep brain areas with high spatial resolution, down to a few cubic millimeters. In this study, the investigators aim to use TUS to non-invasively modulate the globus pallidus internus (GPi) in patients with Parkinson's disease (PD) and dystonia. These patients have previously been implanted with deep brain stimulation (DBS) leads. The investigators plan to simultaneously record local field potentials (LFPs) from the DBS leads using the Percept PC device (Medtronic Inc.) while the DBS is turned off. The study's goal is to investigate the mechanism of action of TUS and its neuromodulatory effects on LFPs recorded from the GPi. This will enable us to compare the effects of TUS with those of DBS.

DETAILED DESCRIPTION:
Study Participants and Visits: The investigators will recruit 10-15 PD and dystonia patients who have undergone DBS with lead locations at the GPi. These participants will be involved in three study visits.

First Visit - MRI Scanning: During the first visit, participants will undergo a structural MRI scan, including T1 and T2 scans, at the Toronto Western Hospital using a 3.0 T Siemens MR-imager. These scans are crucial for transcranial ultrasound modeling to accurately localize the targets.

Second and Third Visits - Transcranial Ultrasound Stimulation (TUS): For the second and third visits, the investigators will use the Brainsight system and BabelBrain, an open source application, to neuronavigate the TUS transducer (NeuroFUS system). This process involves sonication of the GPi, with individualized modeling and simulations to account for ultrasound losses due to variations in skull density and morphology. The investigators will target the GPi bilaterally (where the DBS electrodes are located) and record local field potentials (LFPs) before, during, and up to one hour post TUS.

TUS Protocols: Patients will undergo two different TUS protocols across the recording visits, assigned in random order and spaced at least one week apart. The protocols include:

A tbTUS protocol (5Hz Pulse Repetition Frequency [PRF]), previously shown to increase motor cortex excitability for about one hour after sonication and a 10Hz protocol, which has been demonstrated to inhibit motor cortical activity for about one hour post sonication.

Additionally, the investigators will administer two sham-TUS protocols at each visit, randomly selected to assess placebo effects and the impact of somatosensory stimulation associated with TUS.

The sham protocols are an active sham-TUS for which the investigators will sonicate the occipital cortex (Isppa: 30 W/cm2) using either 5 or 10 Hz protocols, and a passive sham-TUS for which the GPi will be sonicated with either 5 or 10 Hz protocols but at zero power (Isppa: 0 W/cm2).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with movement disorders (diagnosed by a movement disorder specialist)
2. Implantation of a Percept PC DBS system at least one month before the sonications
3. Stable dopaminergic medication dose for a minimum of 4 weeks

Exclusion Criteria:

1. Concomitant neurological conditions (stroke, seizure, dementia, major depression / psychiatric disorders, active drug abuse/addiction and major neuromuscular/musculoskeletal diseases)
2. Declined cognitive scores (MoCA score < 22)
3. Implants (cardiac pacemaker, implantable cardioverter-defibrillator, intracranial devices other than DBS system such as shunts and MR- unsafe devices)
4. History of intracranial lesioning procedures
5. Major systemic illness, infection or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Any treatment-related adverse events and side effects of TUS applications | Two assessments will be conducted during each study visit: one at baseline (within the first minute of the study) and the other upon completion of the study visit (between 150 and 180 minutes after the study visit initiation).
  Adverse effects or side effects, as reported by the neurologist participating throughout the study, will be documented. The neurologist will conduct comprehensive neurological assessments, including cranial nerve evaluations, strength tests, sensory and memory examinations, as well as assessments of coordination and reflexes.
Modulations in the amplitude of the LFP power spectrum | 4-minute long recordings at 1) Baseline (10 minutes before TUS), 2) during TUS (lasting either 120 seconds or 40 seconds, depending on the protocol), 3) 10 minutes after TUS, 4) 30 minutes after TUS, and 5) 45 minutes after TUS
  The power modulations will be measured across different frequencies (theta, alpha, beta) and at different time points (before, during, and after TUS application at each visit).

SECONDARY OUTCOMES:
Modulations of the aperiodic activities derived from the LFPs | 4-minute long recordings at 1) Baseline (10 minutes before TUS), 2) during TUS (lasting either 120 seconds or 40 seconds, depending on the protocol), 3) 10 minutes after TUS, 4) 30 minutes after TUS, and 5) 45 minutes after TUS
  The LFPs will be fitted to classical models of synaptic plasticity. The aperiodic activities derived from the LFPs, along with the results from the synaptic plasticity models, will be compared to investigate the potential mechanisms underlying neuroplasticity induced by TUS.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, MBBS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No